CLINICAL TRIAL: NCT02109692
Title: Quantification of Muscle Specific microRNAs in the Serum of Patients With Duchenne Muscular Dystrophy (DMD) and Becker (BMD) : Evaluation of the Inters-est of These Biomarkers in Patients Care
Brief Title: Evaluation of Muscle miRNA as Biomarkers in Dystrophinopathies
Acronym: biodystromirs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9184
Record Dates: First submitted 2014-04-02; First posted 2014-04-10 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Muscular Dystrophies; Becker Muscular Dystrophy; Duchenne Muscular Dystrophy
Keywords: muscle dystrophies; dystromirs; longitudinal study; miRNA
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cohort (Other): blood sample : doage of miRNA
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — dosage of miRNA

SUMMARY:
Duchenne muscular dystrophy (DMD) , caused by mutations in the DMD gene, is the most common and most severe progressive dystrophy of the child. Although the development is rapidly progressive , there is variability in the severity of the disease between DMD patients that do not correlate with the type of mutations in the DMD gene. There are no easily measurable biomarkers for monitoring the DMD or moderate form of the disease, Becker muscular dystrophy (BMD ) . MicroRNAs (miRNAs) are involved in most cellular processes , and their expression pattern is a signature of the state of a cell . They represent a potential class of diagnostic and prognostic biomarkers. Some are specific for the skeletal myogenesis , and changes in their pattern of expression are associated with muscle diseases including muscular dystrophy. The levels of muscle- specific miRNAs are indeed greatly increased in the serum of DMD and BMD compared to control patients .

The main objective of this is to validate the use of serum muscle-derived microRNAs as biomarkers of DMD patients (compared with healthy subjects). Secondary objectives are i) to investigate the relationship between circulating levels of these miRNAs and the severity of the dystrophinopathy (DMD vs BMD) and also the progression of the disease (longitudinal study), ii) to assess the specificity of these markers for dystrophinopathy (comparison with other patients with muscular dystrophy), iii) to test candidate miRNAs recently identified but not yet analyzed in the serum of patients.

Clinical data and samples will be recorded at each regular consultation. miRNA levels will be quantified using Real Time Quantitative RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from dystrophinopathy or other muscle dystrophy,
* Healthy volunteers
* signed informed consent
* social insurance

Exclusion Criteria:

* patients or parents have not signed the informed consent,

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2014-05-19 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Quantity of serum muscle-derived microRNAs of DMD patients | up to 12 months
  To validate the use of serum muscle-derived microRNAs as biomarkers of DMD patients (compared with healthy subjects)

SECONDARY OUTCOMES:
severity of the dystrophinopathy | up to 36 months
  to investigate the relationship between circulating levels of these miRNAs and the severity of the dystrophinopathy
progression of the disease | up to 36 months
  to investigate the relationship between circulating levels of these miRNAs and the progression of the disease
specificitiy of miRNA for distrophinopathy | up to 36 months
  to assess the specificity of these markers for dystrophinopathy (comparison with other patients with muscular dystrophy)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Rivier, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Montpellier Hospital, Montpellier, France